CLINICAL TRIAL: NCT04396847
Title: Human Laboratory Screening of Lorcaserin in Smokers With Alcohol Use Disorder
Brief Title: Laboratory Screening of Lorcaserin for Alcohol Use Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Medication removed from the U.S. market by the The Food and Drug Administration
Sponsor: The Mind Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 04719
Record Dates: First submitted 2020-02-03; First posted 2020-05-21 (Actual); Results first posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Alcohol Use Disorder; Tobacco Smoking
MeSH Terms: conditions — Alcoholism; Tobacco Smoking | interventions — lorcaserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lorcaserin first, then placebo (Experimental): Participants first receive lorcaserin (10 mg BID) for 7 days. After a washout period of 7 days, they then receive placebo tablets (BID) for 7 days.
  Interventions: Drug: Lorcaserin Oral Tablet
- Placebo first, then lorcaserin (Placebo Comparator): Participants first receive placebo (BID) for 7 days. After a washout period of 7 days, they then receive lorcaserin (10 mg BID) for 7 days.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Lorcaserin Oral Tablet — Lorcasering 10mg Oral Tablet (BID)
  Other Names: Belviq
  Arms: Lorcaserin first, then placebo
Drug: Placebo oral tablet — Placebo Oral Tablet (BID)
  Other Names: Placebo pill
  Arms: Placebo first, then lorcaserin

SUMMARY:
Heavy-drinking smokers, including those with alcohol use disorder (AUD), are at increased risk for numerous negative health outcomes relative to those who use alcohol or cigarettes only. Although heavy-drinking smokers are recognized as an important subgroup for clinical and public health interventions, there are presently no approved medications for the joint indication of alcohol reduction and smoking cessation. Based on evidence that the serotonin system plays a role in alcohol and nicotine consumption and relapse, this study aims to examine whether a serotonin medication alters alcohol and nicotine responses in smokers with AUD, informing its potential utility as a candidate therapy for this clinical subgroup.

DETAILED DESCRIPTION:
Pharmacotherapy development remains a critical objective for reducing health and societal burdens associated with alcohol use disorder (AUD). Developing targeted treatments for specific AUD subgroups is a key objective. Among those with AUD, cigarette smokers comprise a sizable and critical subgroup with disproportionally high long-term health risks, making it a key priority to advance therapies for concurrent AUD and cigarette smoking. The serotonin (5-hydroxtytryptamine; 5-HT) system is broadly implicated in addictive behaviors, in part reflecting the role of 5-HT in modulating dopamine function. Preclinical studies of 5-HT receptor drugs have shown that targeted modulation of the 5-HT2C receptor (implicated in 5-HT-related inhibition of DA function) alters the consumption and reinstatement of addictive drugs, including alcohol and nicotine. Of the selective 5-HT2C receptor agonists, lorcaserin has superior near-term potential for repurposing as an AUD therapy, having been approved by the Food and Drug Administration for weight management. Human laboratory medication trials offer a time- and cost-effective option for validating preclinical findings prior to larger randomized controlled trials, and for testing candidate treatment mechanisms. This Phase II human laboratory screening trial will evaluate lorcaserin as a novel candidate therapy for smokers with AUD. Effects of lorcaserin vs. placebo will be evaluated in a double-blind, within-subjects, crossover study with human laboratory endpoints. This study will provide early human data on the effects of a 5-HT2C receptor agonist in relation to alcohol-related outcomes, informing its potential for further evaluation as a candidate treatment for AUD.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-65
2. Meeting DSM-5 criteria for current (past year) AUD, as well as current at-risk drinking (i.e., ≥14/21 drinks per week for women/men, on average), with at least four episodes of 4+/5+ drinks in the past 30 days
3. Daily smoker, defined as reporting smoking 1+ cigarettes per day, on average, over the past 12 months
4. Willingness to take study pills and complete study procedures
5. Willingness to complete lab sessions involving alcohol administration

Exclusion Criteria:

1. Recent (30 day) illicit drug use (with the exception of cannabis) based on self-report or toxicology screen
2. Meeting DSM-5 criteria for a past-year substance use disorder other than alcohol use disorder, tobacco use disorder, or mild cannabis use disorder
3. Significant alcohol withdrawal, based on a Clinical Institute Withdrawal Assessment for Alcohol-revised (CIWA-Ar) score of 8+ at baseline medical visit, or any reported history of severe withdrawal symptoms (e.g., seizures)
4. Past 30-day use of nicotine replacement
5. Past 30-day use of SSRIs, other psychiatric medications, or weight control medications
6. Lifetime diagnosis of severe mental illness (e.g., psychotic or bipolar I disorder)
7. Significant medical or neurological illness based on medical staff (i.e., physician or nurse practitioner) evaluation including severe hepatic impairment or cirrhosis, insulin dependent diabetes
8. Current alcohol or smoking cessation treatment or efforts to cut down on drinking/smoking
9. Medications contraindicated for use with lorcaserin or which have a significant interaction with lorcaserin
10. Body mass index (BMI) under normal range (<18kg/m2)
11. History of significant cardiovascular conditions including history of arrhythmias or heart block, heart failure, valvular heart disease, heat attack, stroke, unstable angina
12. Abnormal electrocardiogram (ECG) results
13. Currently nursing, pregnant, or anticipating pregnancy
14. history of suicide attempt or recent suicidal ideation (i.e., Suicidal thoughts (intent or plan) in the last month)
15. Plans to travel outside of the local area during the study period, or inability to commit to entire duration of study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 5 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hendershot, Ph.D., Principal Investigator — The Mind Research Network; Eric Claus, Ph.D., Principal Investigator — The Mind Research Network
Locations (1):
- The Mind Research Network, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lorcaserin First, Then Placebo | Placebo First, Then Lorcaserin
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 5 participants provided informed consent. Due to participant no-shows and the cancelation of the study, only one participant started study medication.
Groups:
- Lorcaserin First, Then Placebo: Lorcaserin (10mg BID), then placebo pill (BID)
- Placebo First, Then Lorcaserin: Placebo pill (BID), then Lorcaserin (10mg BID)
- Total: Total of all reporting groups
Arm/Group | Lorcaserin First, Then Placebo | Placebo First, Then Lorcaserin | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Laboratory Alcohol Consumption
Description: Number of drinks consumed during a 2-hour alcohol self-administration session
Time Frame: Laboratory session following 7 days of medication or laboratory session following 7 days of placebo pills.
Population: The trial was halted after randomizing the first two participants. Only one participant completed the dependent measures.
Measure: Number; unit: drinks
Groups:
- Lorcaserin: Lorcaserin (10mg BID)
  Lorcaserin Oral Tablet: Lorcasering 10mg Oral Tablet (BID)
- Placebo: Placebo pill (BID)
  Placebo oral tablet: Placebo Oral Tablet (BID)
Arm/Group | Lorcaserin | Placebo
Number analyzed (Participants) | 1 | 1
drinks | 6 | 4

2. Secondary Outcome: Subjective Responses to Alcohol
Description: Maximum self-reported stimulation during alcohol self-administration, as measured by the Brief Biphasic Alcohol Effects Scale. The final reported score is the sum of each item in the stimulation scale divided by the total number of items (3). The range of scores is 0-10, with higher numbers indicating higher subjective stimulation from alcohol.
Time Frame: Laboratory session following 7 days of medication or laboratory session following 7 days of placebo pills
Population: as for outcome 1
Measure: Number; unit: score on a scale
Arm/Group | Lorcaserin | Placebo
Number analyzed (Participants) | 1 | 1
score on a scale | 3 | .33

3. Secondary Outcome: Motivation to Consume Alcohol
Description: Self-reported alcohol demand, as measured by elasticity in the Alcohol Purchase Task. Elasticity was computed according to Jacobs & Bickel (1999), using the estimated parameters a and b from the equation ln C = ln L + b(ln P) - aP, where C is number of drinks that would be consumed at price P, and L is a constant that represents the number of drinks consumed at P = 1. Overall elasticity is determined by computing elasticity (a-b(P)) for each price/consumption pair and taking the mean. Greater values of elasticity (i.e., less negative in this case) indicate increased willingness to consume the same number of drinks even as the price increases.
Time Frame: Laboratory session following 7 days of medication or laboratory session following 7 days of placebo pills.
Population: as for outcome 1
Measure: Number; unit: elasticity
Arm/Group | Lorcaserin | Placebo
Number analyzed (Participants) | 1 | 1
elasticity | -1.685 | -1.682

4. Secondary Outcome: Motivation to Smoke Cigarettes
Description: Self-reported cigarette demand, as measured by elasticity in the Cigarette Purchase Task. Elasticity was computed according to Jacobs & Bickel (1999), using the estimated parameters a and b from the equation ln C = ln L + b(ln P) - aP, where C is number of cigarettes that would be purchased at price P, and L is a constant that represents the number of cigarettes purchased at P = 1. Overall elasticity is determined by computing elasticity (a-b(P)) for each price/consumption pair and taking the mean. Greater values of elasticity (i.e., less negative in this case) indicate increased willingness to purchase the same number of cigarettes even as the price increases.
Time Frame: Laboratory session following 7 days of medication or laboratory session following 7 days of placebo pills.
Population: as for outcome 1
Measure: Number; unit: elasticity
Arm/Group | Lorcaserin | Placebo
Number analyzed (Participants) | 1 | 1
elasticity | -1.540 | -1.682

5. Secondary Outcome: Daily Alcohol Consumption
Description: Self-reported drinks per drinking day
Time Frame: During 7 days of medication or during 7 days of placebo pills.
Population: as for outcome 1
Measure: Number; unit: Drinks per drinking day
Arm/Group | Lorcaserin | Placebo
Number analyzed (Participants) | 1 | 1
Drinks per drinking day | 10.6 | 11

6. Secondary Outcome: Cigarette Consumption
Description: Number of cigarettes smoked per day
Time Frame: During 7 days of medication or during 7 days of placebo pills.
Population: as for outcome 1
Measure: Number; unit: cigarettes per day
Arm/Group | Lorcaserin | Placebo
Number analyzed (Participants) | 1 | 1
cigarettes per day | 11.4 | 12

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Lorcaserin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT04396847/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT04396847/ICF_001.pdf